CLINICAL TRIAL: NCT00152854
Title: A Randomised, Placebo-controlled, Crossover Trial of Acetaminophen in Cancer Patients on Strong Opioids
Brief Title: Acetaminophen for Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACETAPLAC
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cancer; Pain
Keywords: cancer pain; acetaminophen; opioids
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Acetaminophen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A, 1, acetaminophen (Active Comparator): acetaminophen
  Interventions: Drug: Acetaminophen
- B placebo (Placebo Comparator): placebo PO qid
  Interventions: Drug: placebo, sugar pill

INTERVENTIONS:
Drug: Acetaminophen — acetaminophen 1g po qid
  Arms: A, 1, acetaminophen
Drug: acetaminophen — acetaminophen 1g po qid for 7 days
  Arms: A, 1, acetaminophen
Drug: placebo, sugar pill
  Arms: B placebo

SUMMARY:
Many patients with cancer pain have pain not fully controlled on opioids (eg. morphine). The addition of acetaminophen (Tylenol) to opioids in a small study in cancer patients demonstrated better pain control without an increase in side effects. This study will determine if regular acetaminophen improves pain control when added to strong opioids in patients with cancer pain.

DETAILED DESCRIPTION:
Aim:

To assess whether regular oral acetaminophen can reduce pain in cancer patients already on a strong opioid regimen.

Rationale:

It is estimated that 75% of people with advanced cancer suffer significant pain. Many of these people continue to have pain despite being on strong opioids. The rationale behind adding an additional analgesic with a different mechanism of action is to attempt to improve analgesia without increasing side effects.

Overview:

This is a double blind, randomised placebo-controlled, crossover trial to evaluate whether the addition of regular acetaminophen can reduce pain in cancer patients already on a strong opioid regimen. The study will be performed in ambulatory cancer patients who have pain that is believed to be caused by their cancer, and who have already been stabilised on an opioid regimen of > 60mg/day of morphine equivalents. Each patient will be randomly allocated to receive either acetaminophen 1g qid or an identical appearing placebo qid for a seven-day period, and then crossed over to the other arm for a further seven-day period. Patients will complete daily pain diaries and weekly questionnaires (Brief Pain Inventory) and comparison will be made between the pain scores for the two treatment periods. Patient preference for the two treatment periods will also be evaluated.

Research Question:

A randomised, double-blind, placebo controlled crossover trial to determine if the addition of regular acetaminophen (1g PO qid) leads to improved analgesic control in adult cancer patients at Princess Margaret Hospital, who are already on strong opioids (> 60mg morphine equivalents/day) as evaluated by daily pain scores measured by Numerical Rating Scales (NRS) and the Brief Pain Inventory (BPI).

Hypothesis:

Regular acetaminophen improves pain control in cancer patients who are already on strong opioid regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with malignancy who have persistent pain which is believed by the investigator to be due to their cancer, and whose analgesic regimen has been stabilised on > 60mg of morphine equivalents/day.
2. Age > 18 years
3. Performance status of 0-2 by the European Co-operative Oncology Group (ECOG) Performance Scale
4. Sufficient English skills to be able to complete the daily diary, BPI and to understand the consent form
5. Signed informed consent

Exclusion Criteria:

1. Patient has no pain (0/10 on NRS).
2. Patients with severe pain are excluded, however once their pain control is optimised they are eligible.
3. Patient has received radiation therapy in the six weeks prior to commencing the study or is likely to require radiotherapy during the study period.
4. Patient has commenced, or had dose modifications, to either non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroids in the week prior to commencing the study, or during the two-week study period.
5. Patient has commenced chemotherapy or hormone therapy in the 4 weeks prior to the study or is expected to commence chemotherapy or hormonotherapy during the study period. Patients who are stable on long-term chemotherapy or hormones are eligible for this study. Patients who receive high dose steroids as antiemetics with their chemotherapy are eligible providing they are not receiving the steroids during the study period.
6. Patient has a contraindication to acetaminophen.
7. Use of acetaminophen in the 48 hours prior to commencement of the study period.
8. Abnormal laboratory values:

   * Absolute neutrophil count < 1.5 X 10^9/L and white blood cell (WBC) count < 3 X 10^9/L
   * Platelet count < 100 X 10^9/L
   * Liver transaminases > 2.5 X upper limit of normal
   * Bilirubin > 1.5 X upper limit of normal
   * Creatinine > 1.5 X upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Patient preference for the acetaminophen or the placebo arm as assessed by asking the patient whether he/she preferred treatment period 1 or treatment period 2 | Post completion of period 2
Differences in the mean pain intensity score as assessed by the daily average Numeric Rating Scale (NRS) pain score during the week given acetaminophen compared with the daily average NRS pain score during the week given placebo | post period 2

SECONDARY OUTCOMES:
Symptoms possibly associated with acetaminophen use for each period using an NRS: feeling sick (nausea and vomiting) | post period 2
drowsiness | post period 2
constipation | post period 2
cold sweats | post period 2
overall sense of well being | post period 2
Total analgesic consumption in each treatment period | post period 2
Best and worst pain scores for each treatment period | post period 2
Pain relief obtained in each treatment period | post period 2
Effect of pain on functional ability | post period 2
Strength of preference for acetaminophen versus placebo on a 5-point scale | post period 2
Proportion of patients who had a preference for acetaminophen who perceived the improvement warranted taking the additional tablets | post period 2
Proportion of patients having a clinically significant improvement in pain (defined as an improvement in mean NRS of at least 33% during the week taking acetaminophen) | post period 2

CONTACTS AND LOCATIONS:
Overall Officials: Janette Vardy, MD, Principal Investigator — University Health Network, University of Toronto; David Warr, MD, Principal Investigator — University Health Network, University of Toronto; Ian Tannock, MD, PhD, Principal Investigator — University Health Network, University of Toronto
Locations (2):
- Sydney Cancer Centre, Sydney, New South Wales, Australia
- Princess Margaret Hospital, Toronto, Ontario, Canada